CLINICAL TRIAL: NCT05431725
Title: A Phase Ⅲ, Randomized, Double-blind and Controlled Clinical Trial to Evaluate the Immunogenicity and Safety of Influenza Vaccine (Split Virion), Inactivated, Quadrivalent in Individuals Aged 3 Years and Older
Brief Title: Immunogenicity and Safety Study of Influenza Vaccine (Split Virion), Inactivated, Quadrivalent
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-QINF-3004
Record Dates: First submitted 2022-06-19; First posted 2022-06-24 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Seasonal Influenza
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinovac-QIV group (Experimental): 800 subjects aged 3 years and older will receive one dose of Sinovac-QIV for vaccine-primed subjects or two doses of Sinovac-QIV for vaccine-unprimed subjects.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent
- Vaxigrip Tetra-QIV group (Active Comparator): 800 subjects aged 3 years and older will receive one dose of Vaxigrip Tetra-QIV for vaccine-primed subjects or two doses of Vaxigrip Tetra-QIV for vaccine-unprimed subjects.
  Interventions: Biological: Control Quadrivalent influenza virus vaccine

INTERVENTIONS:
Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent — The influenza vaccines (Split Virion), inactivated, quadrivalent are developed by Sinovac Biotech Co., Ltd.15 μg hemagglutinin (HA) of each of the four influenza strains in 0.5 mL of sodium chloride,disodium hydrogen phosphate, sodium dihydrogen phosphate per injection.The routine of administration is intramuscular injection into deltoid region.
  Other Names: Sinovac-QIV
  Arms: Sinovac-QIV group
Biological: Control Quadrivalent influenza virus vaccine — The Control Quadrivalent influenza virus vaccines are manufactured by Sanofi and are purchased by Pontifical Catholic University of Chile.15μg HA of each of the four influenza strains in 0.5 mL of solution per injection.The routine of administration is intramuscular injection into deltoid region.
  Other Names: Vaxigrip Tetra-QIV
  Arms: Vaxigrip Tetra-QIV group

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of Influenza vaccine (Split virion), Inactivated, Quadrivalent developed by Sinovac Biotech Co., Ltd. (Sinovac-QIV) as compared to a licensed comparator in Chile and Philippines, Vaxigrip Tetra™ (Vaxigrip Tetra-QIV) in individuals aged 3 years and older.

DETAILED DESCRIPTION:
This study is a phase Ⅲ, double-blind, randomized and active-controlled clinical trial to evaluate the safety and immunogenicity of Influenza vaccine (Split virion), Inactivated, Quadrivalent developed by Sinovac Biotech Co., Ltd. (Sinovac-QIV) as compared to a licensed comparator in Chile, Vaxigrip Tetra™ (Vaxigrip Tetra-QIV) in individuals aged 3 years and older. Subjects will be randomized 1:1 to received either Sinovac-QIV or Vaxigrip Tetra-QIV. Vaccine-primed subjects will receive one 0.5ml dose of Sinovac-QIV or Vaxigrip Tetra-QIV on day 0. Vaccine-unprimed subjects will receive two 0.5ml doses of Sinovac-QIV or Vaxigrip Tetra-QIV and day 0 and day 28, respectively. Subjects who are 3-8 years of age had prior receipt of ≥2 doses of influenza vaccine at least 4 weeks apart or who are ≥9 years old are considered "vaccine-prime". Subjects who are 3-8 years of age had prior receipt of <2 dose of influenza vaccine are considered "vaccine-unprimed".

ELIGIBILITY:
Inclusion Criteria:

* Volunteers age 3 years and older, in good health or medically stable;
* Written informed consent obtained from subjects or/and legal guardian;
* No receipt of influenza vaccines within 6 months or plans to receive any influenza vaccines during the study;
* Female subjects of non-child bearing may be enrolled in the study. Non-child bearing potential is defined as surgically sterile (history of bilateral tubal ligation, bilateral oophorectomy, hysterectomy) or premenarche or postmenopausal (defined as amenorrhea for ≥ 12 consecutive months prior to screening without an alternative medical cause);
* Female subjects of child bearing potential may be enrolled in the study, if the subject

  * Has a negative pregnancy test on the day of the first dose (day 0);
  * Has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first dose and until at least 28 days after vaccination.

Exclusion Criteria:

* History of seasonal influenza within 6 months prior to the study entry;
* Axillary temperature ≥37.3℃;
* History of Guillain-Barré syndrome within 6 weeks of receipt of prior influenza vaccine;
* History of allergy to any vaccine, or any ingredient of the experimental vaccine;
* Serious adverse reaction(s) to the vaccine, such as urticaria, dyspnea or angioneurotic edem etc.;
* History of serious neurological disorder (such as epilepsy, convulsions etc.) or a mental illness;
* Autoimmune disease or immunodeficiency/immunosuppressive, or any immunosuppressant receipt within 6 months prior to the study entry;
* Significant chronic illnesses that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion (may include, but are not limited to cardiovascular disease, hypertension and diabetes that cannot be controlled by drugs, liver or kidney disorders, HIV infection or malignant tumor;
* Acute central nervous system diseases such as encephalitis/myelitis, acute disseminating encephalomyelitis, and related disorders;
* Absence of spleen, functional absence of spleen, and absence or removal of spleen under any circumstances;
* Diagnosed coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities), or obvious bruising or coagulation disorders;
* Alcoholism or history of drug abuse；
* Acute disease or acute stage of chronic disease within 7 days prior to study entry;
* Received blood products within 3 months prior to study entry;
* Received any live attenuated vaccine within 14 days prior to study entry or any subunit vaccine or inactivated vaccine within 7 days prior to study entry;
* Pregnant women or lactating women;
* Subjects participate other clinical trials (licensed or unlicensed vaccines, drugs, organisms, devices, blood products or drugs) during the study period;
* Any other factors which are unsuitable for participation in the clinical trial as judged by the investigator.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2202 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates of HI antibody | At day 28 after the last dose
  Seroconversion rates of HI antibody at day 28 after the last dose for each of the four antigens.
GMTs of HI antibody | At day 28 after the last dose
  GMTs of HI antibody at day 28 after the last dose for each of the four antigens.

SECONDARY OUTCOMES:
Seroprotection rates(SCRs) of HI antibody | At day 28 after the last dose
  Proportion of subjects with antibody titer ≥1:40 at day 28 after the last dose
Seroconversion rates (SCRs) of HI antibody | At day 28 after the last dose
  Seroconversion rates at day 28 after the last dose.
Solicited local and systemic Adverse Events (AEs) | Within 7 days after each dose
  Occurrence, intensity, duration, and relationship of solicited local and systemic Adverse Events (AEs) within 7 days after each dose.
Unsolicited AEs | Within 28 days after each dose
  Occurrence, intensity, duration, and relationship of unsolicited AEs within 28 days after each dose.
Serious adverse events (SAEs) | Within 28 days after each dose
  Occurrence and relationship of serious adverse events (SAEs) within 28 days after each dose
Adverse events of special interest (AESI) | Within 28 days after each dose
  Adverse events of special interest (AESI) within 28 days after each dose

CONTACTS AND LOCATIONS:
Overall Officials: Zeng Gang, Senior Medical Director, Study Director — Sinovac Biotech Co., Ltd
Locations (11):
- Chile (7):
  - Hospital de Puerto Montt, Port Montt
  - CIMER Center/Center for Medical Research on Respiratory Diseases, Santiago
  - Clínica Alemana, Santiago
  - Hospital Clínico UC-Christus, Santiago
  - Hospital Felix Bulnes, Santiago
  - Universidad San Sebastián, Santiago
  - Clinica Alemana de Valdivia, Valdivia
- Philippines (4):
  - Las Pinas Doctors Hospital, Las Piñas, Manila
  - Tropical Disease Foundation Inc, Makati City, Manila
  - San Juan De Dios Hospital, Pasay, Manila
  - Philippine General Hospital, Manila